CLINICAL TRIAL: NCT03875417
Title: Multidisciplinary HCC Treatment in Elderly : QoL and Survival Analysis
Brief Title: Multidisciplinary Management of HCC in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Professor Stefania Brozzetti, Associate Professor, Azienda Policlinico Umberto I
Other Study IDs: HEP001
Record Dates: First submitted 2019-03-10; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: HCC; Quality of Life
Keywords: HCC; HCC in elderly; recurrent HCC; Liver resection; Quality of Life; intervention radiology; RF; TACE
MeSH Terms: interventions — Hepatectomy; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients who developed HCC recurrences after surgery and treated with re-resection, or microinvasive non-surgical means.
  Interventions: Procedure: liver resection; Procedure: Thermic ablation; Procedure: Transcatheter arterial chemoembolization
- Group B: Patients who did not develop recurrences after surgery.
  Interventions: Procedure: liver resection

INTERVENTIONS:
Procedure: liver resection — resection of one or more HCC nodules within the liver
Procedure: Thermic ablation — ablation of HCC nodule through a percutaneous needle, by using radiofrequency or microwaves
  Other Names: RF (radiofrequency ablation) / MWA (microwaves ablation)
  Groups: Group A
Procedure: Transcatheter arterial chemoembolization — embolization of HCC nodule via drug-eluted microbeads.
  Groups: Group A

SUMMARY:
Aim of this study is to evaluate whether treating HCC recurrences in resected elderly patients is advantageous or not.

DETAILED DESCRIPTION:
Introduction- Hepatocellular carcinoma (HCC) is the most common primary liver malignancy. It usually develops in cirrhotic liver with high recurrence rates. More than 2/3 of patients are elderly, often excluded from surgery and follow-up protocols. Aim of this study is to evaluate whether treating HCC recurrences in resected elderly patients is advantageous or not.

Materials and methods- 126 patients, aged between 65 and 90 years, submitted to liver resection for HCC were enrolled. They were divided into three classes. Class 1 included patients submitted to major resections, Class 2 to minor resections and Class 3 to minor resections associated with thermoablation. All of them were clinically and radiologically followed up. Patients who developed recurrences (Group A) were referred to further treatments (surgery, interventional radiology or pharmacological therapy). Mortality, disease-free survival (DFS), overall survival (OS) and quality of life (QoL) were evaluated and compared with non-recurrent patients (Group B).

Used interventional radiology means were Radiofrequency ablation (RF), microwaves ablation (MWA) or transcatheter arterial chemoembolization (TACE).

ELIGIBILITY:
Inclusion Criteria:

* HCC patient
* eligible for surgery

Exclusion Criteria:

* non eligible for surgery at first HCC diagnosis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: all patients submitted to surgery for HCC nodules resection between 2002 and 2017
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | follow up time 1-16 years
  survival in months
Disease free survival | follow up time 1-16 years
  survival without recurrences in months

SECONDARY OUTCOMES:
Karnofsky performance scale | follow up time 1-16 years
  evaluation of performance status in dimensionless scale 0 - 100
Activity of Daily living | follow up time 1-16 years
  assess the ability to manage common routine activities evaluated in dimensionless scale 1-6
Instrumental Activity of Daily living | follow up time 1-16 years
  assess the ability to use common instruments evaluated in dimensionless scale 1-8
Blood Haemoglobin | follow up time 1-16 years
  evaluation of mean haemoglobin levels in g/dl
serum Albumin | follow up time 1-16 years
  evaluation of mean albumin levels in g/dl
Geriatric Depression Scale | follow up time 1-16 years
  evaluation of depression in patients in dimensionless scale 0 - 15

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Brozzetti, Professor, Principal Investigator — Policlinico Umberto I - Sapienza università di Roma
Locations (1):
- Department of Surgery "Pietro Valdoni", Roma, Italy

IPD SHARING:
Plan to Share IPD: No